CLINICAL TRIAL: NCT05115032
Title: Randomized Controlled Trial of Computerized Dynamic Posturography-assisted Vestibular Retraining Compared With At-home Vestibular Rehabilitation Exercises for Stable Unilateral Vestibular Deficit
Brief Title: Posturography-assisted Vestibular Retraining for Stable Unilateral Vestibular Deficit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eytan A. David (Other)
Responsible Party: Sponsor-Investigator, Eytan A. David, MD, FRCSC, Clinical Instructor, Dept. of Surgery, University of British Columbia
Organization: University of British Columbia (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: H21-03343
Record Dates: First submitted 2021-10-29; First posted 2021-11-10 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2024-05

CONDITIONS: Dizziness; Equilibrium; Disorder, Labyrinth; Inner Ear Injury; Inner Ear Disease
MeSH Terms: conditions — Dizziness; Labyrinth Diseases

STUDY DESIGN:
Intervention Model Description: Randomized controlled interventional trial; single crossover; single-centre, open label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Vestibular retraining with dynamic posturography (Experimental): 12 sessions, twice per week, of rehabilitation exercises last about 20 minutes, using CDP and interactive visual feedback
  Interventions: Device: Vestibular retraining with dynamic posturography
- At-home rehabilitation exercises (Active Comparator): Daily rehabilitation exercises involving nodding and shaking of the head
  Interventions: Behavioral: At-home rehabilitation exercises

INTERVENTIONS:
Device: Vestibular retraining with dynamic posturography — 12 sessions, twice per week, of rehabilitation exercises last about 20 minutes, using CDP and interactive visual feedback
  Arms: Vestibular retraining with dynamic posturography
Behavioral: At-home rehabilitation exercises — 6 weeks of daily rehabilitation exercises involving nodding and shaking of the head
  Arms: At-home rehabilitation exercises

SUMMARY:
People that have difficulty with balance have a higher risk of falling and reduced quality of life. Some individuals can learn to compensate using their vision, their sense of where their limbs are in space, and balance organs that are still intact. Rehabilitation exercises, which typically involve shaking and nodding of the head, are often prescribed for dizzy patients but are not effective for everyone. Our study aims to determine if specific exercises performed on footplate sensors with visual feedback is superior to traditional rehabilitation exercises done at home for improving balance and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Dizziness handicap inventory score at time of enrolment over 30
* Unilateral vestibular weakness confirmed one or more of:

  * Videonystagmography showing unilateral weakness to bithermal testing of greater than 25%
  * VEMP: IAD asymmetry of greater than 40% for both cVEMP and oVEMP
  * VEMP: absence of both ocular and cervical vemp responses in one ear in the context of normal and replicable other ear
  * Or unilateral vestibular weakness idiopathic, not yet diagnosed (NYD)
* Persistent imbalance following diagnosis of resolved benign paroxysmal positional vertigo (BPPV)
* Symptomatic
* Long-standing/persistent symptoms greater than six months

Exclusion Criteria:

* Orthopedic deficit (eg. lower body joint dysfunction or lower joint replacement)
* Neurological deficit or proprioception deficit
* Diabetes
* Poor vision or blindness
* Fluctuating vestibular symptoms, or condition known to fluctuate eg. Menière's disease, perilymphatic fistula (PLF) or superior canal dehiscence (SDCS)
* Active benign paroxysmal positional vertigo (BPPV)
* Undergoing treatment which may affect balance or ability to stand
* Cognitive impairment that prevents understanding and responding to instructions required to complete the study
* Inability to provide informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2022-01-17 (Actual); Primary Completion 2022-12-15 (Actual); Study Completion 2023-04-19 (Actual)

PRIMARY OUTCOMES:
SOT composite score | Through study completion, 12 rehabilitation sessions, an average of 7 weeks
  Change in composite score of sensory organization test (Scores from 0-100; higher scores indicate better function)
Dizziness Handicap Inventory | Through study completion, 12 rehabilitation sessions, an average of 7 weeks
  Change in Dizziness Handicap Inventory (DHI); 16-30 Points (mild handicap), 32-52 Points (moderate handicap), 54+ Points (severe handicap)

SECONDARY OUTCOMES:
ABC Score | Through study completion, 12 rehabilitation sessions, an average of 7 weeks
  Change in Activity-specific Balance Confidence (ABC) score; (Scores from 0-100; higher scores indicate better function)
FES-I score | Through study completion, 12 rehabilitation sessions, an average of 7 weeks
  Change in Fall Efficacy Scale-International (FES-I); possible scores 16-64, higher score indicates greater impairment
SOT condition scores | Through study completion, 12 rehabilitation sessions, an average of 7 weeks
  Change in mean SOT scores for conditions 1 through 6; (Scores from 0-100; higher scores indicate better function)
LOS directional control | Through study completion, 12 rehabilitation sessions, an average of 7 weeks
  Limits of Stability test mean value of directional control of limits of stability; (Scores from 0-100; higher scores indicate better function)
LOS excursion | Through study completion, 12 rehabilitation sessions, an average of 7 weeks
  Limits of Stability test mean endpoint excursion value and maximum excursion point; (Scores from 0-100; higher scores indicate better function)
DHI component scores | Through study completion, 12 rehabilitation sessions, an average of 7 weeks
  Emotional, physical, and functional components of the DHI score
SOT vestibular contribution | Through study completion, 12 rehabilitation sessions, an average of 7 weeks
  Change in mean value of SOT condition 5/mean value of SOT conditions 1; measured as a ratio, higher scores indicate a greater vestibular contribution to balance deficit

CONTACTS AND LOCATIONS:
Overall Officials: Eytan A David, MD, Principal Investigator — University of British Columbia
Locations (1):
- Dr. EA David MD FRCSC, North Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] David EA, Shahnaz N, Wiseman I, David Y, Cochrane CL. Vestibular Rehabilitation Using Dynamic Posturography: Functional Stability and Fall Risk Outcomes From a Randomized Trial. Otolaryngol Head Neck Surg. 2025 Sep;173(3):713-723. doi: 10.1002/ohn.1302. Epub 2025 Jul 7. PMID 40624853